CLINICAL TRIAL: NCT01762982
Title: A Single Centre, Examiner-blind Human Patch Test of Bactroban Disinfectant Liquid on Normal Skin
Brief Title: Patch Test of Benzalkonium Chloride Disinfectant Spray
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RH01379
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-07

CONDITIONS: Wound Healing
MeSH Terms: interventions — Benzalkonium Compounds; sodium lactobionate sucrose solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test (Experimental): Benzalkonium chloride (0.13%) Disinfectant Spray water
  Interventions: Drug: 0.13% Benzalkonium Chloride
- Positive Control (Active Comparator): Sodium lauryl sulfate (SLS) (0.3% weight by weight [w/w]) water solution
  Interventions: Drug: SLS Solution
- Negative Control 1 (Placebo Comparator): Normal saline water (0.9% weight by volume [w/v])
  Interventions: Drug: Normal Saline Water
- Negative Control 2 (Placebo Comparator): Empty Finn Chamber
  Interventions: Other: Empty Finn Chamber

INTERVENTIONS:
Drug: 0.13% Benzalkonium Chloride — Finn Chamber filled with benzalkonium chloride (0.13%) disinfectant spray water solution
  Arms: Test
Drug: SLS Solution — Finn Chamber filled with SLS (0.3% w/v) water solution
  Arms: Positive Control
Drug: Normal Saline Water — Finn Chamber filled with Normal Saline water (0.9% w/v)
  Arms: Negative Control 1
Other: Empty Finn Chamber — Empty Finn Chamber
  Arms: Negative Control 2

SUMMARY:
The aim of the study is to evaluate the irritation potential of benzalkonium chloride disinfectant spray when placed in contact with normal human skin.

DETAILED DESCRIPTION:
Benzalkonium chloride is recognized as safe and effective for short term use as first aid antiseptic drug products. In this study, benzalkonium chloride disinfectant spray will be compared to a positive control, and two negative control for irritancy potential on normal skin according to Chinese Patch Test Guideline (China Health Authority 2002). The skin irritation assessment will characterize the test products individually in terms of symptomatology using a 5-point categorical scale ranging from 0 (no visible reaction) to 4 (Erythema,edema˛ extreme blistering).

ELIGIBILITY:
Inclusion Criteria:

1. Consent: Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
2. Compliance: Understands and is willing, able and likely to comply with all study procedures and restrictions, and will agree to not participate in any other study during the entire length of the study.
3. General Health: Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history and vital signs at the screening.
4. Contraception: Females of childbearing potential who are, in the opinion of the investigator, practising a reliable method of contraception.

Exclusion Criteria:

1. Pregnancy: Woman who is pregnant or who has a positive urine pregnancy test (just for females of childbearing potential) at the baseline.
2. Breast-feeding: Woman who is breast-feeding.
3. Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials or have self-reported "sensitive skin" or a history of dermal hypersensitivity.
4. Clinical Study/Experimental Medication: Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit, including those who have taken part in any predictive irritation study or sensitisation test.
5. Substance abuse: Recent history (within the last 1 year) of alcohol or other substance abuse.
6. Personnel: An employee of the sponsor or the study site or members of their immediate family.
7. Participant who is currently taking any of the following medications:

   * Any topical or systemic treatments that may mask or interfere with the test results, specifically topical and/or systemic corticosteroids, non steroidal anti-inflammatory drugs (e.g. ibuprofen, aspirin), antihistamines and immunosuppressive in the past 30 days. And those taking medications which in the opinion of the clinical investigator may affect test results.
   * Topical anti-inflammation treatment in the aimed application area in the past 2 months.
8. Participant who has a history of any acute or chronic disease that might interfere with or increase the risk on study participation. (e.g., atopic dermatitis/eczema, systemic lupus erythematosus, rheumatoid arthritis, other autoimmune diseases, asthma and other chronic respiratory disease).

10. Participant who has damaged skin in close proximity to test sites (e.g., sunburn, uneven skin pigmentation, tattoos, scars, birthmarks or other disfigurations). And those who are suffering from any active skin disorders, conditions, or any visible skin disease which might be confused with a skin reaction from the test materials.

11. Participant who requires use of any emollient on the upper back throughout the study or who use of any emollient or other skin care product on the upper back in the past 3 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- PeKing University First Hospital, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Of 37 participants screened, 1 did not meet the study criteria. Remaining 36 were randomized to the study. Two negative controls, one positive control and one test product were used simultaneously and inserted into the patch (Finn chamber patch test device) as it was a 4-way split plot design study.
Groups:
- Overall: This was a 4-way split-plot clinical study. Four Finn chambers which contained the test product (Benzalkonium chloride solution; 0.03 milliliters (mL) of 0.13% Benazalkonium chloride solution), one positive control [Sodium lauryl sulphate (SLS); 0.03 mL of 0.3% weight by weight (w/w) SLS solution] and 2 negative controls including one chamber for normal saline (0.03 mL of 0.9% weight by volume (w/v) normal saline) and an empty Finn chamber were applied on the left upper back of each subject for 24 hours under occlusive dressing. The sequence of the patch assembly (Finn chambers) was randomized. During this 24 hour patch applications, subjects had direct and ongoing skin contact with the investigational products and the positive and negative controls.
Period: Overall Study
Arm/Group | Overall
Started | 36
Received Saline Water | 36
Received Benzalkonium Chloride | 36
Received SLS | 36
Received Empty Finn Chamber | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were evaluated for baseline parameters.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.2 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Skin Irritation Scores at 24 Hours
Description: Irritation potential of the treatments was assessed by proportion of the irritation scores by a trained dermatologist. Skin Irritation reaction was categorized as: 0=No visible reaction; 1= Weak Erythema (Redness); 2=Erythema, Infiltration, Papule; 3= Erythema, Edema, Papule, Blister; 4=Erythema, Edema, Extreme Blistering. For the product to be deemed as non-irritant to skin, requirements were proportion of score of 2 should not be more than 1 out of 15 participants and no cases of score of 3 or 4.
Time Frame: Baseline to 24 hours following product application
Population: Intention to Treat (ITT) population: All randomized participants who received the study treatments at baseline and had at least one post baseline skin irritation scoring assessment.
Measure: Number; unit: Percentage of participants
Groups:
- Benzalkonium Chloride Solution: 0.03 mL of 0.13% Benazalkonium chloride solution, filled in a Finn chamber was applied to upper back of participants for 24 hours.
- SLS Solution: 0.03 mL of 0.3% w/w SLS solution, filled in a Finn chamber was applied to upper back of participants for 24 hours.
- Normal Saline Water: 0.03 mL of 0.9% w/v normal saline, filled in a Finn chamber was applied to upper back of participants for 24 hours.
- Empty Finn Chamber: Empty Finn Chamber (a patch test device) was applied to upper back of participants for 24 hours.
Arm/Group | Benzalkonium Chloride Solution | SLS Solution | Normal Saline Water | Empty Finn Chamber
Number analyzed (Participants) | 36 | 36 | 36 | 36
Percentage of participants
  Score = 0 (No Visible Skin Reaction) | 75.0 | 91.7 | 94.4 | 94.4
  Score = 1 (Weak Erythema) | 25.0 | 8.3 | 5.6 | 5.6
  Score = 2 (Erythema, Infiltration, Papule) | 0 | 0 | 0 | 0
  Score = 3 (Erythema, Edema, Papule, Blister) | 0 | 0 | 0 | 0
  Score = 4 (Erythema, Edema, Extreme Blistering) | 0 | 0 | 0 | 0

2. Secondary Outcome: Skin Irritation Scores at 24 Hours
Description: as for outcome 1
Time Frame: Baseline to 24 hours following product application
Population: ITT population: All randomized participants who received the study treatments at baseline and had at least one post baseline skin irritation scoring assessment. Missing data was not imputed.
Measure: Number; unit: Number of participants
Arm/Group | Benzalkonium Chloride Solution | Normal Saline Water
Number analyzed (Participants) | 36 | 36
Number of participants
  Score = 0 (No Visible Skin Reaction) | 27 | 24
  Score = 1 (Weak Erythema) | 9 | 2
  Score = 2 (Erythema, Infiltration, Papule) | 0 | 0
  Score = 3 (Erythema, Edema, Papule, Blister) | 0 | 0
  Score = 4 (Erythema, Edema, Extreme Blistering) | 0 | 0
Statistical Analysis 1: Comparison: Benzalkonium Chloride Solution vs Normal Saline Water; Null hypothesis considered no treatment difference between the treatments being compared; Test type: Superiority or Other; p = 0.0654, Signed Rank Test; Median Difference (Final Values) = 0.0

3. Primary Outcome: Proportion of Participants With Skin Irritation Scores at 48 Hours
Description: as for outcome 1
Time Frame: Baseline to 48 hours following first product application
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Benzalkonium Chloride Solution | SLS Solution | Normal Saline Water | Empty Finn Chamber
Number analyzed (Participants) | 36 | 36 | 36 | 36
Percentage of participants
  Score = 0 (No Visible Skin Reaction) | 77.8 | 50.0 | 100.0 | 100.0
  Score = 1 (Weak Erythema) | 22.2 | 38.9 | 0 | 0
  Score = 2 (Erythema, Infiltration, Papule) | 0 | 11.1 | 0 | 0
  Score = 3 (Erythema, Edema, Papule, Blister) | 0 | 0 | 0 | 0
  Score = 4 (Erythema, Edema, Extreme Blistering) | 0 | 0 | 0 | 0

4. Primary Outcome: Proportion of Participants With Skin Irritation Scores at 72 Hours
Description: as for outcome 1
Time Frame: Baseline to 72 hours following first product application
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Benzalkonium Chloride Solution | SLS Solution | Normal Saline Water | Empty Finn Chamber
Number analyzed (Participants) | 36 | 36 | 36 | 36
Percentage of participants
  Score = 0 (No Visible Skin Reaction) | 77.8 | 61.1 | 94.4 | 100.0
  Score = 1 (Weak Erythema) | 16.7 | 22.2 | 5.6 | 0
  Score = 2 (Erythema, Infiltration, Papule) | 5.6 | 16.7 | 0 | 0
  Score = 3 (Erythema, Edema, Papule, Blister) | 0 | 0 | 0 | 0
  Score = 4 (Erythema, Edema, Extreme Blistering) | 0 | 0 | 0 | 0

5. Secondary Outcome: Skin Irritation Scores at 48 Hours
Description: as for outcome 1
Time Frame: Baseline to 48 hours following first product application
Population: as for outcome 2
Measure: Number; unit: Number of participants
Arm/Group | Benzalkonium Chloride Solution | Normal Saline Water
Number analyzed (Participants) | 36 | 36
Number of participants
  Score = 0 (No Visible Skin Reaction) | 28 | 36
  Score = 1 (Weak Erythema) | 8 | 0
  Score = 2 (Erythema, Infiltration, Papule) | 0 | 0
  Score = 3 (Erythema, Edema, Papule, Blister) | 0 | 0
  Score = 4 (Erythema, Edema, Extreme Blistering) | 0 | 0
Statistical Analysis 1: Comparison: Benzalkonium Chloride Solution vs Normal Saline Water; Null hypothesis considered no treatment difference between the treatments being compared; Test type: Superiority or Other; p = 0.0078, Signed Rank Test; Median Difference (Final Values) = 0.0

6. Secondary Outcome: Skin Irritation Scores at 72 Hours
Description: as for outcome 1
Time Frame: Baseline to 72 hours following first product application
Population: as for outcome 2
Measure: Number; unit: Number of participants
Arm/Group | Benzalkonium Chloride Solution | Normal Saline Water
Number analyzed (Participants) | 36 | 36
Number of participants
  Score = 0 (No Visible Skin Reaction) | 28 | 34
  Score = 1 (Weak Erythema) | 6 | 2
  Score = 2 (Erythema, Infiltration, Papule) | 2 | 0
  Score = 3 (Erythema, Edema, Papule, Blister) | 0 | 0
  Score = 4 (Erythema, Edema, Extreme Blistering) | 0 | 0
Statistical Analysis 1: Comparison: Benzalkonium Chloride Solution vs Normal Saline Water; Null hypothesis considered no treatment difference between the treatments being compared; Test type: Superiority or Other; p = 0.0547, Signed Rank Test; Median Difference (Final Values) = 0.0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the start of the investigational product and until 5 days following last administration of the investigational product.
Description: This was a 4 way Split-plot design study. Hence, all the treatments were given at the same time so association of any adverse event with one specific treatment was not justifiable.
Groups:
- Overall Study: This was a 4-way split-plot study. Four Finn chambers which contained the test product (Benzalkonium chloride solution; 0.03 mL of 0.13% Benazalkonium chloride solution), one positive control [SLS; 0.03 mL of 0.3% w/w SLS solution] and 2 negative controls including one chamber for normal saline (0.03 mL of 0.9% w/v normal saline) and an empty Finn chamber were applied on the left upper back of each subject for 24 hours under occlusive dressing. The sequence of the patch assembly (Finn chambers) was randomized. During this 24 hour patch applications, subjects had direct and ongoing skin contact with the investigational products and the positive and negative controls.
  All randomized participants exposed to at least one of the study treatments were evaluated for safety.
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 3/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=36)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.